CLINICAL TRIAL: NCT07233005
Title: The Effect of Quadriceps Sets Exercise on Knee Joint Biomechanics and Functional Outcomes of Post-Total Knee Arthroplasty Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rokaia Ali Zainelabedeen Mohamed Toson, Assistant Professor of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-03-46
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadriceps Set & Terminal Knee Extension Exercises Group (Study Group) (Experimental)
  Interventions: Procedure: Quadriceps Set Exercise; Procedure: Terminal Knee Extension; Procedure: Traditional Physical Therapy
- Traditional Physical Therapy Group (Control Group) (Experimental)
  Interventions: Procedure: Traditional Physical Therapy

INTERVENTIONS:
Procedure: Quadriceps Set Exercise — Quadriceps knee set exercises was introduced with the patient in sitting position and pillow was placed under his knee joint then ask patient to dorsiflex his ankle and extend knee make hold 10 second then relax. Two exercises session per week for four week.
  Arms: Quadriceps Set & Terminal Knee Extension Exercises Group (Study Group)
Procedure: Terminal Knee Extension — Terminal knee extension exercise using Thera band was introduced with the patient in sitting or standing position and the theraband was placed around his knee joint. Two exercises session per week for four week.
  Arms: Quadriceps Set & Terminal Knee Extension Exercises Group (Study Group)
Procedure: Traditional Physical Therapy — Traditional physical therapy program will include passive stretching exercise to the hamstrings while the patient is supine lying flex the hip while the knee extended and hold for 30-45 seconds, strengthening exercise to the guadriceps muscle by extending the knee whie the patient is in the sitting position.

SUMMARY:
Lower limb strengthening, especially the quadriceps training, is of much necessity for patients with knee arthroplasty. As the quadriceps strengthening exercises play a vital role in controlling gait pattern during walking and different activities. Vastus inetrmedius muscle responsible for the last 10 degree of knee extension. This enable the knee joint to be in locked position which is the stable position during gait.

ELIGIBILITY:
Inclusion Criteria:

1. Age (ranging from 40 to 60 years old).
2. Weight (ranging from 65 to 75 kg).
3. Height (ranging from 150 to 165 cm)
4. Sex ( male/ female).
5. Patients who undergoing total knee arthroplasty after 1 months until one year after operation.

Exclusion Criteria:

1. Cognitive impairment.
2. Neuromuscular impairment.
3. Patient can't walk alone (need of assistive device).

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analoge Scale (VAS) | Four weeks
  VAS is a straight horizontal line of usually 100 mm. The ends are defined as the extreme limits of the pain . It is orientated from the left (worst) to the right (least) pain.
Quadriceps Muscle Strength | 4 weeks
  it will be measured using a hand held dynamometer.

SECONDARY OUTCOMES:
Range of Motion (ROM) | 4 weeks
  ROM of last ten degree of knee extension measured by goniometer
Oxford Knee Score (OKS) | 4 weeks
  The OKS is a patient reported outcome measure that consists of 12 questions about an individual's level of function, activities of daily living and how they have been affected by pain over the preceding four weeks.The Oxford Knee Score (OKS) ranges from 0 to 48, 0 = Worst possible knee pain/function. 48 = Best possible knee pain/function.
The Western Ontario and McMaster Universities Osteoarthritis Index (The WOMAC) | 4 weeks
  It is a questionnaire of 24-item. Self-administered tool used to assess pain, stiffness, and physical function in patients with hip and knee osteoarthritis.
  WOMAC Likert Version (0-96 total)
  Each item scored:
  0 = none
  1. = mild
  2. = moderate
  3. = severe
  4. = extreme Total score ranges from: 0 = best possible (no symptoms). 96 = worst possible (severe symptoms).

CONTACTS AND LOCATIONS:
Locations (1):
- Jouf University, Sakakah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes